CLINICAL TRIAL: NCT03151993
Title: Multicenter Open Label Randomized Comparative Study of Efficacy and Safety of Single Bolus Injection of Recombinant Nonimmunogenic Staphylokinase (Fortelyzin) and Bolus Infusion Alteplase (Actilyse) in Patients With Acute Ischemic Stroke
Brief Title: Single Bolus Recombinant Nonimmunogenic Staphylokinase (Fortelyzin) and Bolus Infusion Alteplase in Patients With AIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supergene, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRIDA Stroke Trial
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke
Keywords: Acute Ischemic Stroke; Fibrinolysis; Fortelyzin
MeSH Terms: conditions — Ischemic Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: All eligible patients will be randomized in two equal groups for administration recombinant nonimmunogenic staphylokinase (Fortelyzin) or alteplase (Actilyse) by using "envelope method" of randomization. It is an open-lable study. Each of agents will be administered no longer then 4,5 hours from symptoms onset. Comparative agent will be administered as prescribed in its instructions. All patients will be examination for 90 days
Masking Description: All eligible patients will be randomized in two equal groups for administration recombinant nonimmunogenic staphylokinase (Fortelyzin) or alteplase (Actilyse) by using "envelope method" of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant staphylokinase (Experimental): Lyophilizate for solution making for intravenous injection, 5 mg (745000 ME). 10 mg of drug reconstituted in 10 ml of 0.9% solution of NaCl given as single i.v. bolus over 5 - 10 seconds
  Interventions: Drug: Recombinant staphylokinase
- Actilyse (Active Comparator): Intravenous alteplase 0.9 mg/kg (10% bolus and 90% as IV infusion over 1 hour, maximum 90 mg)
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Recombinant staphylokinase — 10 mg of drug reconstituted in 10 ml of 0.9% solution of NaCl given as single i.v. bolus over 5 - 10 seconds
  Other Names: Fortelyzin
  Arms: Recombinant staphylokinase
Drug: Alteplase — Intravenous alteplase 0.9 mg/kg (10% bolus and 90% as IV infusion over 1 hour, maximum 90 mg)
  Other Names: Actilyse
  Arms: Actilyse

SUMMARY:
The aim of the study is to determine if single-bolus recombinant nonimmunogenic staphylokinase is effective and save thrombolytic agent in patients with ischemic stroke in comparison to alteplase.

DETAILED DESCRIPTION:
Experimental Drug Profile. The active substance of Fortelyzin is Forteplase. It's recombinant protein which contains aminoacid sequence of staphylokinase. It is single chain molecula, consists of 138 aminoacids, weight 15.5 kDa. When staphylokinase is added to human plasma containing a fibrin clot, it preferentially reacts with plasmin at the clot surface, forming a plasmin-staphylokinase complex. This complex activates plasminogen trapped in the thrombus. The plasmin-staphylokinase complex and plasmin bound to fibrin are protected from inhibition by alpha2-antiplasmin. Once liberated from the clot (or generated in plasma), however, they are rapidly inhibited by alpha2-antiplasmin. This selectivity of action confines the process of plasminogen activation to the thrombus, preventing excessive plasmin generation, alpha2-antiplasmin depletion, and fibrinogen degradation in plasma. In rabbits anti forteplase antibodies are not produced. It was achieved by replacement of amino acids in immunogenic epitop of molecule staphylokinase. Blood fibrinogen decrease after i.v. injection of Fortelyzin less 10% within first 24 hours. Angiographic data suggests that restoration of coronary blood flow appears in up to 80% of patients with STEMI after i.v. injection of Fortelyzin.

Main goals of the study are to prove an efficacy of the single-bolus intravenous injection of recombinant nonimmunogenic staphylokinase (Fortelyzin) in comparison with bolus infusion alteplase(Actilyse) in patients with ischemic stroke.

To prove a safety and to assess possible adverse events in the single-bolus intravenous injection of recombinant nonimmunogenic staphylokinase (Fortelyzin) in comparison with bolus infusion alteplase (Actilyse) in patients with ischemic stroke.

Study Design. All eligible patients will be randomized in two equal groups for administration recombinant nonimmunogenic staphylokinase (Fortelyzin) or alteplase (Actilyse) by using "envelope method" of randomization. It is an open-lable study. Each of agents will be administered no longer then 4,5 hours from symptoms onset. Comparative agent will be administered as prescribed in its instructions. All patients will be examination for 90 days

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 80 (Version 1.0)
* Men and women aged 18 years and older, after 80 years with caution (Version 2.0)
* Verified diagnosis of ischemic stroke (from 5 to 25 points on the NIHSS scale). (Version 1.0)
* Verified diagnosis of ischemic stroke (Version 2.0)
* The time from the onset of the disease is no more than 4.5 hours.
* Informed consent received

Exclusion Criteria:

* The time of the onset of the first symptoms is more than 4.5 hours from the onset of the disease or the time of the onset of the first symptoms of a stroke is not known (for example, the development of a stroke during sleep - the so-called "night stroke").
* Increased sensitivity to alteplase, gentamicin (residual traces from the production process).
* Systolic blood pressure above 185 mm Hg. Art. Or diastolic blood pressure above 110 mm Hg. Art. Or the need for / in the administration of drugs to reduce blood pressure to these boundaries.
* Neuroimaging (CT, MRI) signs of intracranial hemorrhage, brain tumors, arteriovenous malformation, brain abscess, aneurysm of cerebral vessels.
* Surgery on the brain or spinal cord.
* Suspicion of subarachnoid hemorrhage.
* Signs of severe stroke: clinical signs (stroke scale NIH> 25), neuroimaging (according to CT of the brain and / or MRI of the brain in the DWI, the ischemia focuses on the territory of more than 1/3 of the CMA pool).
* Simultaneous reception of oral anticoagulants, for example, warfarin with INR> 1.3.
* The use of direct anticoagulants (heparin, heparinoids) in the preceding stroke of 48 h with APTT values above the norm.
* Prior stroke or severe head injury within 3 months.
* Significant regression of neurological symptoms during the observation of the patient.(Version 1.0)
* Light neurological symptoms (NIH <4 points). (Version 1.0)
* Significant regression of neurological symptoms during the observation of the patient before thrombolisis (Version 2.0)
* Hemorrhagic stroke or stroke, unspecified in history.
* Strokes of any genesis in the history of a patient with diabetes mellitus.
* Gastrointestinal bleeding or bleeding from the genitourinary system in the last 3 weeks. Confirmed exacerbations of gastric ulcer and duodenal ulcer during the last 3 months.
* Extensive bleeding now or within the previous 6 months.
* Severe liver disease, including liver failure, cirrhosis, portal hypertension (with varicose veins of the esophagus), active hepatitis.
* Acute pancreatitis.
* Bacterial endocarditis, pericarditis.
* Aneurysms of arteries, malformations of arteries and veins. Suspicion of exfoliating aortic aneurysm.
* Neoplasms with an increased risk of bleeding.
* Large operations or severe injuries within the last 14 days, minor surgery or invasive manipulation in the last 10 days.
* Puncture of uncompensated arteries and veins during the last 7 days.
* Prolonged or traumatic cardiopulmonary resuscitation (more than 2 min).
* Pregnancy, obstetrics, 10 days after birth.
* The number of platelets is less than 100,000 / μL.
* Blood glucose less than 2.7 mmol / l or more than 22.0 mmol / l.
* Hemorrhagic diathesis, including renal and hepatic insufficiency.
* Data on bleeding or acute trauma (fracture) at the time of examination.
* Seizures in the onset of the disease, if there is no certainty that the seizure is a clinical manifestation of ischemic stroke with a postictal residual deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2017-03-18 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evgenii I Gusev, MD, PhD, Principal Investigator — Pirogov Russian National Research Medical University; Sergey S Markin, MD, PhD, Study Director — Supergene, LLC
Locations (18):
- Russia (18):
  - Regional Clinical Hospital, Barnaul
  - St.Iosaf's Belgorod Regional Clinical Hospital, Belgorod
  - Regional Clinical Hospital №3, Chelyabinsk
  - Regional Clinical Hospital, Irkutsk
  - Regional Clinical Hospital, Kaluga
  - Ochapowski Regional Hospital №1, Krasnodar
  - Regional Clinical Hospital, Kursk
  - Regional Clinical Hospital, Nizhny Novgorod
  - Regional Clinical Hospital, Orenburg
  - City Clinical Hospital №11, Ryazan
  - Regional Clinical Hospital, Ryazan
  - Regional Clinical Hospital, Saint Petersburg
  - Regional Clinical Hospital, Samara
  - Regional Clinical Hospital, Tver'
  - Regional Clinical Hospital, Ulyanovsk
  - City Clinical Hospital of Emergency №25, Volgograd
  - Regional Clinical Hospital №1, Voronezh
  - Regional Clinical Hospital №1, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong PW, Gershlick A, Goldstein P, Wilcox R, Danays T, Bluhmki E, Van de Werf F; STREAM Steering Committee. The Strategic Reperfusion Early After Myocardial Infarction (STREAM) study. Am Heart J. 2010 Jul;160(1):30-35.e1. doi: 10.1016/j.ahj.2010.04.007. PMID 20598969
- [Background] Van de Werf F, Cannon CP, Luyten A, Houbracken K, McCabe CH, Berioli S, Bluhmki E, Sarelin H, Wang-Clow F, Fox NL, Braunwald E. Safety assessment of single-bolus administration of TNK tissue-plasminogen activator in acute myocardial infarction: the ASSENT-1 trial. The ASSENT-1 Investigators. Am Heart J. 1999 May;137(5):786-91. doi: 10.1016/s0002-8703(99)70400-x. PMID 10220625
- [Background] Assessment of the Safety and Efficacy of a New Thrombolytic (ASSENT-2) Investigators; Van De Werf F, Adgey J, Ardissino D, Armstrong PW, Aylward P, Barbash G, Betriu A, Binbrek AS, Califf R, Diaz R, Fanebust R, Fox K, Granger C, Heikkila J, Husted S, Jansky P, Langer A, Lupi E, Maseri A, Meyer J, Mlczoch J, Mocceti D, Myburgh D, Oto A, Paolasso E, Pehrsson K, Seabra-Gomes R, Soares-Piegas L, Sugrue D, Tendera M, Topol E, Toutouzas P, Vahanian A, Verheugt F, Wallentin L, White H. Single-bolus tenecteplase compared with front-loaded alteplase in acute myocardial infarction: the ASSENT-2 double-blind randomised trial. Lancet. 1999 Aug 28;354(9180):716-22. doi: 10.1016/s0140-6736(99)07403-6. PMID 10475182
- [Background] Assessment of the Safety and Efficacy of a New Thrombolytic Regimen (ASSENT)-3 Investigators. Efficacy and safety of tenecteplase in combination with enoxaparin, abciximab, or unfractionated heparin: the ASSENT-3 randomised trial in acute myocardial infarction. Lancet. 2001 Aug 25;358(9282):605-13. doi: 10.1016/S0140-6736(01)05775-0. PMID 11530146
- [Background] Wallentin L, Goldstein P, Armstrong PW, Granger CB, Adgey AA, Arntz HR, Bogaerts K, Danays T, Lindahl B, Makijarvi M, Verheugt F, Van de Werf F. Efficacy and safety of tenecteplase in combination with the low-molecular-weight heparin enoxaparin or unfractionated heparin in the prehospital setting: the Assessment of the Safety and Efficacy of a New Thrombolytic Regimen (ASSENT)-3 PLUS randomized trial in acute myocardial infarction. Circulation. 2003 Jul 15;108(2):135-42. doi: 10.1161/01.CIR.0000081659.72985.A8. Epub 2003 Jul 7. PMID 12847070
- [Background] Vanderschueren S, Dens J, Kerdsinchai P, Desmet W, Vrolix M, De Man F, Van den Heuvel P, Hermans L, Collen D, Van de Werf F. Randomized coronary patency trial of double-bolus recombinant staphylokinase versus front-loaded alteplase in acute myocardial infarction. Am Heart J. 1997 Aug;134(2 Pt 1):213-9. doi: 10.1016/s0002-8703(97)70127-3. PMID 9313600
- [Background] Collaborative Research Group of Reperfusion Therapy in Acute Myocardial Infarction. [A randomized multicenter trial comparing recombinant staphylokinase with recombinant tissue-type plasminogen activator in patients with acute myocardial infarction]. Zhonghua Xin Xue Guan Bing Za Zhi. 2007 Aug;35(8):691-6. Chinese. PMID 17963623
- [Background] Collen D. Staphylokinase: a potent, uniquely fibrin-selective thrombolytic agent. Nat Med. 1998 Mar;4(3):279-84. doi: 10.1038/nm0398-279. No abstract available. PMID 9500599
- [Background] Wahlgren N, Ahmed N, Eriksson N, Aichner F, Bluhmki E, Davalos A, Erila T, Ford GA, Grond M, Hacke W, Hennerici MG, Kaste M, Kohrmann M, Larrue V, Lees KR, Machnig T, Roine RO, Toni D, Vanhooren G; Safe Implementation of Thrombolysis in Stroke-MOnitoring STudy Investigators. Multivariable analysis of outcome predictors and adjustment of main outcome results to baseline data profile in randomized controlled trials: Safe Implementation of Thrombolysis in Stroke-MOnitoring STudy (SITS-MOST). Stroke. 2008 Dec;39(12):3316-22. doi: 10.1161/STROKEAHA.107.510768. Epub 2008 Oct 16. PMID 18927461
- [Background] Hacke W, Kaste M, Fieschi C, von Kummer R, Davalos A, Meier D, Larrue V, Bluhmki E, Davis S, Donnan G, Schneider D, Diez-Tejedor E, Trouillas P. Randomised double-blind placebo-controlled trial of thrombolytic therapy with intravenous alteplase in acute ischaemic stroke (ECASS II). Second European-Australasian Acute Stroke Study Investigators. Lancet. 1998 Oct 17;352(9136):1245-51. doi: 10.1016/s0140-6736(98)08020-9. PMID 9788453
- [Background] Clark WM, Wissman S, Albers GW, Jhamandas JH, Madden KP, Hamilton S. Recombinant tissue-type plasminogen activator (Alteplase) for ischemic stroke 3 to 5 hours after symptom onset. The ATLANTIS Study: a randomized controlled trial. Alteplase Thrombolysis for Acute Noninterventional Therapy in Ischemic Stroke. JAMA. 1999 Dec 1;282(21):2019-26. doi: 10.1001/jama.282.21.2019. PMID 10591384
- [Background] Hacke W, Kaste M, Bluhmki E, Brozman M, Davalos A, Guidetti D, Larrue V, Lees KR, Medeghri Z, Machnig T, Schneider D, von Kummer R, Wahlgren N, Toni D; ECASS Investigators. Thrombolysis with alteplase 3 to 4.5 hours after acute ischemic stroke. N Engl J Med. 2008 Sep 25;359(13):1317-29. doi: 10.1056/NEJMoa0804656. PMID 18815396
- [Derived] Gusev EI, Martynov MY, Nikonov AA, Shamalov NA, Semenov MP, Gerasimets EA, Yarovaya EB, Semenov AM, Archakov AI, Markin SS; FRIDA Study Group. Non-immunogenic recombinant staphylokinase versus alteplase for patients with acute ischaemic stroke 4.5 h after symptom onset in Russia (FRIDA): a randomised, open label, multicentre, parallel-group, non-inferiority trial. Lancet Neurol. 2021 Sep;20(9):721-728. doi: 10.1016/S1474-4422(21)00210-6. PMID 34418399
- See also: Efficacy Guidelines. The work carried out by ICH under the Efficacy heading is concerned with the design, conduct, safety and reporting of clinical trials. — http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Recombinant Staphylokinase | Actilyse
Started | 168 | 168
Completed | 168 | 168
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recombinant Staphylokinase | Actilyse | Total
Number analyzed (Participants) | 168 | 168 | 336
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 84 | 80 | 164
  >=65 years | 84 | 88 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (9.6) | 64.6 (10.6) | 64.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 112 | 218
  Male | 62 | 56 | 118
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 168 | 168 | 336
Baseline NIHSS score [Median (Inter-Quartile Range); unit: score] — The median of The National Institutes of Health Stroke Scale (NIHSS), where: 0 - No stroke symptoms, 1-4 - Minor stroke, 5-15 - Moderate stroke, 16-20 - Moderate to severe stroke, 21-42 - Severe stroke.
  score | 11 [8 to 14] | 11 [8 to 16] | 11 [8 to 15]
Baseline mRS score [Median (Inter-Quartile Range); unit: score] — The median of The Modified Rankin Scale (mRS): 0 - No symptoms, 1 - No significant disability. All scale is 0 - No symptoms, 1 - No significant disability, 2 - Slight disability, 3 - Moderate disability, 4 - Moderately severe disability, 5 - Severe disability, 6 - Dead.
  score | 4 [4 to 5] | 4 [4 to 5] | 4 [4 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Good Functional Recovery
Description: The number of patients with Modified Rankin Scale (mRS) scores 0-1 on day 90 after drug administration, where 0 - No symptoms, 1 - No significant disability. All scale is 0 - No symptoms, 1 - No significant disability, 2 - Slight disability, 3 - Moderate disability, 4 - Moderately severe disability, 5 - Severe disability, 6 - Dead.
Time Frame: within 90 days after fibrinolysis
Measure: Number; unit: patients
Arm/Group | Recombinant Staphylokinase | Actilyse
Number analyzed (Participants) | 168 | 168
patients | 84 | 68
Statistical Analysis 1: Comparison: Recombinant Staphylokinase vs Actilyse; Test type: Non-Inferiority — The non-inferiority hypothesis would be declared if the lower limit of the 95% CI for an mRS score of 0-1 on day 90 did not cross the margin of noninferiority of 16%. The non-inferiority hypothesis was tested using Welch's t-test for the primary outcome only; p < 0.01, Welch's t-test; Odds Ratio (OR) = 9.5, 95% CI 2-sided [-1.7 to 20.7]

2. Secondary Outcome: The Number of Patients With Modified Rankin Scale (0-1) + NIHSS (0-1) + Barthel (95-100)
Description: Composite endpoint, included the number of patients reached Modified Rankin scale 0-1 score, NIHSS 0-1 score and Barthel index 95-100.
  Modified Rankin scale: 0 - No symptoms, 1 - No significant disability, 2 - Slight disability, 3 - Moderate disability, 4 - Moderately severe disability, 5 - Severe disability, 6 - Dead.
  The National Institutes of Health Stroke Scale (NIHSS): 0 - No stroke symptoms, 1-4 - Minor stroke, 5-15 - Moderate stroke, 16-20 - Moderate to severe stroke, 21-42 - Severe stroke.
  Barthel index: 80-100 - Independent, 60-79 - Minimally dependent, 40-59 - Partially dependent, 20-39 - Very dependent, <20 - Totally dependent.
Time Frame: within 90 days after fibrinolysis
Measure: Number; unit: patients
Arm/Group | Recombinant Staphylokinase | Actilyse
Number analyzed (Participants) | 168 | 168
patients | 59 | 52

3. Secondary Outcome: The Median of NIHSS After 24 Hours
Description: The median of The National Institutes of Health Stroke Scale (NIHSS) at 24 h after drug administration, where: 0 - No stroke symptoms, 1-4 - Minor stroke, 5-15 - Moderate stroke, 16-20 - Moderate to severe stroke, 21-42 - Severe stroke.
Time Frame: after 24 hours
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | Recombinant Staphylokinase | Actilyse
Number analyzed (Participants) | 168 | 168
score | 6 [3 to 11] | 6 [3 to 12]

4. Secondary Outcome: The Median of NIHSS After 90 Days
Description: The median of The National Institutes of Health Stroke Scale (NIHSS) after 90 days of drug administration, where: 0 - No stroke symptoms, 1-4 - Minor stroke, 5-15 - Moderate stroke, 16-20 - Moderate to severe stroke, 21-42 - Severe stroke.
Time Frame: within 90 days after fibrinolysis
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | Recombinant Staphylokinase | Actilyse
Number analyzed (Participants) | 168 | 168
score | 2 [1 to 5] | 2 [1 to 5]

5. Secondary Outcome: All Cause Death
Description: Death caused by any event
Time Frame: within 90 days after fibrinolysis
Measure: Number; unit: patients
Arm/Group | Recombinant Staphylokinase | Actilyse
Number analyzed (Participants) | 168 | 168
patients | 17 | 24

6. Secondary Outcome: Intracranial Haemorrhage
Description: The number of intracranial hemorrhage (events)
Time Frame: within 90 days after fibrinolysis
Measure: Number; unit: events
Arm/Group | Recombinant Staphylokinase | Actilyse
Number analyzed (Participants) | 168 | 168
events | 31 | 28

7. Secondary Outcome: Symptomatic Intracranial Haemorrhage
Description: The number of symptomatic intracranial haemorrhage according to ECASS III definition (events). The ECASS III definition of symptomatic intracranial haemorrhage was any haemorrhage with neurologic deterioration, as indicated by an NIHSS score that was higher by 4 points or more than the value at baseline or the lowest value in the first 7 days, or any haemorrhage leading to death. In addition, the haemorrhage must have been identified as the predominant cause of the neurologic deterioration.
Time Frame: within 90 days after fibrinolysis
Measure: Number; unit: events
Arm/Group | Recombinant Staphylokinase | Actilyse
Number analyzed (Participants) | 168 | 168
events | 5 | 13

ADVERSE EVENTS:
Time Frame: 90 days after fibronolysis
Description: Cerebral oedema, Symptomatic intracranial haemorrhage, Surgery, Neurosurgery, Acute myocardial infarction, Pulmonary thromboembolism, New acute ischaemic stroke, Gastric ulcer, Takotsubo cardiomyopathy.
Arm/Group | Recombinant Staphylokinase | Actilyse
All-Cause Mortality (participants affected / at risk) | 17/168 | 24/168
Serious Adverse Events (participants affected / at risk) | 22/168 | 38/168
Other Adverse Events (participants affected / at risk) | 7/168 | 8/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Staphylokinase (N=168) | Actilyse (N=168)
Cerebral oedema (Nervous system disorders) | 7 (7) | 14 (14)
Symptomatic intracranial haemorrhage (Nervous system disorders) | 5 (5) | 13 (13)
Surgery (Nervous system disorders) | 5 (5) | 3 (3)
Neurosurgery (Nervous system disorders) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Pulmonary thromboembolism (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
New acute ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Takotsubo cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Staphylokinase (N=168) | Actilyse (N=168)
Haematuria (Renal and urinary disorders) | 7 (7) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT03151993/Prot_SAP_000.pdf